CLINICAL TRIAL: NCT04959175
Title: Phase I/II Study to Reduce Post-transplantation Cyclophosphamide Dosing for Older or Unfit Patients Undergoing Bone Marrow Transplantation for Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000359; 000359-C
Record Dates: First submitted 2021-07-10; First posted 2021-07-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-12

CONDITIONS: Hematologic Neoplasms
Keywords: myeloablative conditioning; Chronic Graft-Versus-Host Disease; hematopoietic cell transplantation; Fludarabine; TOTAL BODY IRRADIATION
MeSH Terms: conditions — Hematologic Neoplasms; Bronchiolitis Obliterans Syndrome | interventions — Mycophenolic Acid; fludarabine; Sirolimus; Filgrastim; Cyclophosphamide; Mesna; Whole-Body Irradiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Donors (No Intervention): Collection of research samples on bone marrow donors
- Older, HLA-matched (Experimental): Subjects age 60-85 with hematologic malignancies and an HLA-matched related or unrelated donor
  Interventions: Drug: Mycophenolate Mofetil; Procedure: Allogeneic HSCT; Drug: Fludarabine; Drug: Sirolimus; Drug: Filgrastim; Drug: Cyclophosphamide; Drug: Mesna; Procedure: Total Body Irradiation (TBI)
- Older, HLA-mismatched (Experimental): Subjects age 60-85 with hematologic malignancies and an HLA-haploidentical or HLA-mismatched unrelated donor
  Interventions: Drug: Mycophenolate Mofetil; Procedure: Allogeneic HSCT; Drug: Fludarabine; Drug: Sirolimus; Drug: Filgrastim; Drug: Cyclophosphamide; Drug: Mesna; Procedure: Total Body Irradiation (TBI)
- Younger, HLA-matched (Experimental): Subjects age 18-60 unfit for MAC with hematologic malignancies and an HLA-matched related or unrelated donor
  Interventions: Drug: Mycophenolate Mofetil; Procedure: Allogeneic HSCT; Drug: Fludarabine; Drug: Sirolimus; Drug: Filgrastim; Drug: Cyclophosphamide; Drug: Mesna; Procedure: Total Body Irradiation (TBI)
- Younger, HLA-mismatched (Experimental): Subjects age 18-60 unfit for MAC with hematologic malignancies and an HLA-haploidentical or HLA-mismatched unrelated donor
  Interventions: Drug: Mycophenolate Mofetil; Procedure: Allogeneic HSCT; Drug: Fludarabine; Drug: Sirolimus; Drug: Filgrastim; Drug: Cyclophosphamide; Drug: Mesna; Procedure: Total Body Irradiation (TBI)

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 15 mg/kg orally or IV three times daily (max 1000 mg/dose) starting on day +5, continued through day +35. May be continued beyond the protocol specified stop date if there is GVHD or mixed chimerism.
  Arms: Older, HLA-matched; Older, HLA-mismatched; Younger, HLA-matched; Younger, HLA-mismatched
Procedure: Allogeneic HSCT — Stem cell transplant
  Arms: Older, HLA-matched; Older, HLA-mismatched; Younger, HLA-matched; Younger, HLA-mismatched
Drug: Fludarabine — 30 mg/m2 IV infusion over 30-60 minutes once daily for 5 days (Pre-Transplant days -6 through -2).
  Arms: Older, HLA-matched; Older, HLA-mismatched; Younger, HLA-matched; Younger, HLA-mismatched
Drug: Sirolimus — Loading dose of 6 mg orally given on day +5 (calculated based on actual body weight, max initial dose 6 mg), then maintenance dose starting at 2 mg orally daily on day +6 with dose adjustments to maintain a trough of 5-12 ng/ml, continued through day +60 with no taper. May be continued beyond the protocol specified stop date if there is GVHD or mixed chimerism.
  Arms: Older, HLA-matched; Older, HLA-mismatched; Younger, HLA-matched; Younger, HLA-mismatched
Drug: Filgrastim — begins on day +5 at a dose of 5 mcg/kg/day (actual body weight) IV or subcutaneously, until the absolute neutrophil count is > 1,000/mm3 over the course of three days or > 5,000/mm3 on one day. Rounding to the nearest vial is allowed. G-CSF may be stopped early or not administered if required by the clinical circumstance. Additional G-CSF may be administered as warranted.
  Arms: Older, HLA-matched; Older, HLA-mismatched; Younger, HLA-matched; Younger, HLA-mismatched
Drug: Cyclophosphamide — Pre-transplant: 14.5 mg/kg/day IV daily for 2 days pre-transplant (Pre-Transplant days -6 and -5). Post-transplant: 25 mg/kg/day or 35 mg/kg/day (Post-transplant days +3 and +4).
  Arms: Older, HLA-matched; Older, HLA-mismatched; Younger, HLA-matched; Younger, HLA-mismatched
Drug: Mesna — 25 or 35 mg/kg (equal to the cyclophosphamide dose) as IV infusion concomitant with cyclophosphamide. Mesna may or may not be given with the pre-transplant cyclophosphamide depending on institutional practice.
  Arms: Older, HLA-matched; Older, HLA-mismatched; Younger, HLA-matched; Younger, HLA-mismatched
Procedure: Total Body Irradiation (TBI) — 400 centigray (cGy) to be delivered in 2 fractions as 200 cGy per fraction twice daily. Pre-Transplant Day -1 (or Day 0 prior to graft administration)
  Arms: Older, HLA-matched; Older, HLA-mismatched; Younger, HLA-matched; Younger, HLA-mismatched

SUMMARY:
Background:

Certain blood cancers can be treated with blood or bone marrow transplants. Sometimes the donor cells attack the recipient's body, called graft-versus-host disease (GVHD). The chemotherapy drug cyclophosphamide helps reduce the risk and severity of GVHD. Researchers want to learn if using a lower dose of cyclophosphamide may reduce the drug's side effects while maintaining its effectiveness. Such an approach is being used in an ongoing clinical study at the NIH with promising results, but this approach has not been tested for transplants using lower doses of chemotherapy/radiation prior to the transplant.

Objective:

To learn if using a lower dose of cyclophosphamide will help people have a successful transplant and have fewer problems and side effects.

Eligibility:

Adults ages 18-85 who have a blood cancer that did not respond well to standard treatments or is at high risk for relapse without transplant, and their donors.

Design:

Participants may be screened with the following:

Medical history

Physical exam

Blood and urine tests

Heart and lung tests

Body imaging scans (they may get a contrast agent)

Spinal tap

Bone marrow biopsy

Participants will be hospitalized for 4-6 weeks. They will have a central venous catheter placed in a chest or neck vein. It will be used to give medicines, transfusions, and the donor cells, and to take blood. In the week before transplant, they will get 2 chemotherapy drugs and radiation. After the transplant, they will get the study drug for 2 days. They will take other drugs for up to 2 months.

Participants must stay near NIH for 3 months after discharge for weekly study visits. Then they will have visits every 3-12 months until 5 years after transplant.

Participants and donors will give blood, bone marrow, saliva, cheek swab, urine, and stool samples for research.

DETAILED DESCRIPTION:
Background:

With novel therapies for hematologic malignancies, an increasing number of older and/or less fit patients are achieving remissions, but these new therapies are not curative, making consolidation approaches with curative intent such as allogeneic transplantation necessary.

Frailty is a phenotype that predicts a patient s intolerance of physiologic stressors and may predict a patient s tolerance of intensive consolidative strategies.

Frailty phenotype, though increasing in incidence in older patients, can occur in younger patients and may predict poor survival after allogeneic transplantation.

We have yet to define the ideal allogeneic transplantation regimen for older patients or those with frailty or pre-frail phenotypes.

Post-transplantation cyclophosphamide (PTCy) reduces rates of severe acute and chronic graft-versus-host disease (GVHD) after allogeneic hematopoietic cell transplantation (HCT) and safely facilitates human leukocyte antigen (HLA)-matched-related, HLA-matched-unrelated, HLA-mismatched-unrelated, and HLA-haploidentical HCT; it has become the most widely adopted change to transplantation platforms over the last decade.

When clinically translated, the dose (50 mg/kg/day) of PTCy used was partly extrapolated from murine major histocompatibility complex (MHC)-matched skin allografting models and was partly empirical.

In both MHC-haploidentical and MHC-disparate murine HCT models, a dose of 25 mg/kg/day was superior to 50 mg/kg/day on days +3 and +4 in terms of GVHD severity and mortality. Lower dosing of PTCy also was associated with less broad reductions of T-cell numbers after PTCy and lower toxicity than higher dosing.

In patients on an NIH study using myeloablative conditioning, a dose of 25 mg/kg/day has been associated with more rapid engraftment and potentially better immune function without an increase in severe acute GVHD.

Objectives:

Determine whether PTCy 25 mg/kg on days +3 and +4 can maintain adequate protection against grade III-IV acute GVHD and reduce toxicity associated with transplantation in older and/or unfit transplant recipients receiving reduced intensity conditioned allogeneic HCT.

Determine the frailty measures associated with outcomes after allogeneic transplantation.

Eligibility:

Histologically or cytologically confirmed hematologic malignancy with standard indication for allogeneic hematopoietic cell transplantation.

Age 60-85 years, or age 18-60 years and unfit for myeloablative conditioning (MAC).

At least one potentially suitable HLA-matched related, HLA-haploidentical donor, HLA-matched unrelated, or >=5/10 HLA-mismatched unrelated donor.

Karnofsky performance score >=60

Adequate organ function

Design:

Open-label, multi-center, non-randomized, phase I/II study

There will be four separate arms: HLA-matched elderly, HLA-matched young/infirm, HLA-partially matched elderly, and HLA-partially matched young/infirm

All subjects will receive nonmyeloablative conditioning consisting of fludarabine, cyclophosphamide, and total body irradiation; GVHD prophylaxis with PTCy 25 mg/kg on days +3 and +4, MMF, and sirolimus; and bone marrow as the stem cell source

Subjects will be evaluated for development of grade III-IV acute GVHD (aGVHD) at day +60 as the dose-limiting toxicities for the Simon two-stage design. Dose escalation of PTCy will be permitted within each arm if stopping rules are met at the 25 mg/kg/day on days +3 and +4 dose.

Frailty assessments will be performed prior to transplantation conditioning and serially after allogeneic transplantation.

ELIGIBILITY:
-INCLUSION CRITERIA - Recipient

1. Subjects must have a histologically or cytologically confirmed hematologic malignancy with standard indication for allogeneic hematopoietic cell transplantation including, but not limited to, one of the following:

   * Acute myeloid leukemia in morphologic complete remission (<5% blasts in the bone marrow, no detectable abnormal peripheral blasts, and no extramedullary disease)
   * B-cell acute lymphoblastic leukemia in first or subsequent complete remission
   * T-cell acute lymphoblastic leukemia in first or subsequent complete remission
   * Myelodysplastic syndrome of intermediate or higher score by the Revised International Prognostic Scoring System (IPSS-R)
   * Primary myelofibrosis of intermediate-2 or higher risk by the DIPSS
   * Chronic myelomonocytic leukemia
   * Chronic myelogenous leukemia resistant to or intolerant of >=3 tyrosine kinase inhibitors or with history of accelerated phase or blast crisis
   * B-cell lymphoma including Hodgkin lymphoma that has relapsed within 1 year of completion of primary treatment, after autologous transplantation or has progressed through at least 2 lines of therapy
   * Chronic lymphocytic leukemia with 17p deletion and/or unmutated IgHV or refractory or intolerant of both BTK and PI3K inhibitors
   * Mature T or NK neoplasms as defined in the WHO guidelines of sufficient type and severity for allogeneic HCT based on the Prognostic Index for T-cell lymphoma (PIT) score of low-intermediate risk or higher60 or on recently published clinical practice guidelines
   * Hematologic malignancy of dendritic cell or histiocytic cell type
   * Multiple myeloma, stage III, relapsing after therapy with both a proteasome inhibitor and an immunomodulatory drug (IMiD)
2. Age 60-85 years, or age 18-60 years and unfit for myeloablative conditioning. Reasons for unfitness for myeloablative conditioning include:

   * Prior myeloablative HCT
   * Prior exposure to inotuzumab, gemtuzumab, or other agent that increases the risk for sinusoidal obstruction syndrome.
   * Significant organ dysfunction (e.g., creatinine or liver enzymes above the upper limit of normal or EGFR <=70 ml/min/1.73sq.m; prior sinusoidal obstruction syndrome, hepatic fibrosis, hepatic steatosis, or nodular regenerative hyperplasia; reduced ejection fraction <55% or focal hypokinesis, FEV1 or adjusted DLCO <75% of predicted)
   * Hematopoietic Cell Transplantation- Comorbidity Index (HCT-CI) >= 3
   * Subject refusal of MAC (including subjects insistent on trying to maintain fertility)
   * Pre-frail or frail by Fried s frailty phenotype
   * Karnofsky performance score <80
   * Significant life-threatening toxicities associated with prior chemotherapy
   * Co-morbidity considered by the treating physician to be exclusionary of MAC
3. At least one potentially suitable HLA-matched related, HLA-haploidentical first degree or collateral related, HLA-matched unrelated, or >=5/10 HLA-mismatched unrelated donor.
4. Karnofsky performance score >=60
5. Ability of subject to understand and the willingness to sign a written informed consent document.
6. Adequate organ function defined as possessing all of the following:

   * Cardiac ejection fraction >=35%;
   * Forced expiratory volume-1, forced vital capacity, and diffusing capacity of the lung for carbon monoxide (corrected for hemoglobin) all of >=40% predicted;
   * Serum creatinine clearance of >=45 ml/minute calculated using the Cockcroft-Gault equation;
   * Total bilirubin <=2X the upper limit of normal;
   * Alanine aminotransferase and aspartate aminotransferase <=5X the upper limit of normal.
7. Nonmyeloablative conditioning is toxic to the developing human fetus and is teratogenic. For this reason, the following measures apply:

   * Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one year post-transplant.
   * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
   * WOCBP must have a negative serum or urine pregnancy test within 7 days prior to enrollment.
8. For NIH treated subjects only: subjects requiring standard therapies to prepare for HCT should be referred in remission, if possible. However, these diseases are often aggressive and require swift evaluation for HCT while concurrently attempting to establish disease control through the administration of standard therapies. If ongoing therapy for the underlying disease outside of the NIH is not in the best interest of the subject according to the clinical judgment of the NIH PI, then the subject may receive standard treatment for his/her underlying hematologic malignancy as a bridge to HCT on this protocol, prior to starting the research phase of the study. If it becomes apparent that the subject will not be able to proceed to HCT, then he/she must come off study. Subjects receiving standard therapy will be told about the therapy, associated risks, potential benefits, alternatives to the proposed therapy, and the availability of receiving the same treatment elsewhere, outside of a research protocol.

EXCLUSION CRITERIA - Recipient:

1. Subjects who are receiving any other investigational agents. Prior experimental therapies must have been completed at least 2 weeks prior to the date of beginning conditioning.
2. Poorly controlled malignant indication for transplantation such as:

   * Leukemia not having achieved morphologic remission (i.e. bone marrow blasts >5% or active extramedullary disease)
   * Lymphoma not having achieved at least a partial response to prior chemotherapy or radiation
3. Uncontrolled intercurrent illness that in the opinion of the site PI would make it unsafe to proceed with transplantation.
4. The potential for some of the study medications to be transmissible via breast milk of nursing mothers is unknown. Because there is unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding must be discontinued.
5. Active malignancy of non-hematopoietic type which is: metastatic, relapsed/refractory to treatment, or locally advanced and not amenable to curative treatment, or limited disease treated with curative intent treatment within the last 2 years. This excludes nonmelanoma skin cancers.

INCLUSION CRITERIA - Donor:

Related (age >=12) and unrelated (age >=18) donors deemed eligible (i.e., evaluated at NIH in accordance with existing institutional Standard Policies and Procedures or evaluated per the standards required by the IRB of the National Marrow Donor Program or applicable registry), and willing to donate research samples will be included.

EXCLUSION CRITERIA - Donor:

None

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
determine if optimal dose of PTCy to prevent grade III-IV acute GVHD (aGVHD) at day +60 | 60 days
  The fraction of evaluable patients who experience grade III-IV aGVHD at day +60 will be determined and reported along with 80% and 95% two-sided confidence intervals. In addition, a cumulative incidence curve for this endpoint will be constructed.

SECONDARY OUTCOMES:
Grade III-IV acute GVHD at day 100 and 200 | 100 days/200 days
  Estimates will be determined using competing risk-based cumulative incidence curves. Graft failure, relapse, donor lymphocyte infusion, non-relapse mortality, and chronic GVHD will be competing risks for acute GVHD. Grade III-IV aGVHD also will be evaluated descriptively including fractions who attain each condition at day 100 and 200 days, and 95% confidence intervals.
Grade II-IV acute GVHD at day 100 and 200 | 100 days/200 days
  Estimates will be determined using competing risk-based cumulative incidence curves. Grade II-IV aGVHD also will be evaluated descriptively including fractions who attain each condition at day 100 and 200 days, and 95% confidence intervals.
Rate of Fried s Frailty Phenotypes (FP) | 1 year
  Frequency of different phenotypes
Chronic GVHD at one year | 1 year
  Estimates will be determined using competing risk-based cumulative incidence curves. Graft failure, relapse, donor lymphocyte infusion, and non-relapse mortality will be competing risks for chronic GVHD.
Progression/relapse at one year | 1 year
  Estimates will be determined using Kaplan-Meier curves. Relapse and non-relapse mortality will be competing risks for each other.
Non-relapse mortality at 100 days and one year | 100 days and 1 year
  Estimates will be determined using competing risk-based cumulative incidence curves. Relapse and non-relapse mortality will be competing risks for each other.
Overall survival, progression-free survival, and disease-free survival at one year | 1 year
  Estimates will be determined using Kaplan-Meier curves.
Estimation of platelet engraftment, neutrophil engraftment. | day 28 and day 100
  Rate and timing will be evaluated descriptively, including fractions who attain each condition at day 28 and 100, along with 95% confidence intervals. Ranges and medians will be calculated only in engrafting participants.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Kanakry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. @@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000359-C.html